CLINICAL TRIAL: NCT00472810
Title: Comparative Study of the Safety and Effectiveness Between Ologen (OculusGen) Collagen Matrix Implant and Mitomycin-C in Glaucoma Filtering Surgery
Brief Title: Ologen (OculusGen)-Glaucoma MMC Control in Pakistan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pro Top & Mediking Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mediking 0703; OculusGen-2006-02-20
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Glaucoma; Trabeculectomy
Keywords: Glaucoma; Collagen matrix; ologen; OculusGen; Antifibrotic; Trabeculectomy; anti scarring; tissue engineering; high risk patient for trabeculectomy; Aeon Astron
MeSH Terms: conditions — Glaucoma | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 20 patients will be recruited according to the enrollment acceptance criteria.Randomisation is performed using a sealed envelope system, where 40 shuffled envelopes designating the surgery to either trabeculectomy with mitomycin-C (MMC) and trabeculectomy with ologen™ Collagen matrix must be open before surgery. Then, patients are allocated and trabeculectomy is performed.If ologen™ treatment is used, the collagen matrix will be placed on top of the scleral flap under the conjunctiva after the trabeculectomy.
  Interventions: Device: ologen collagen matrix in glaucoma filtering surgery
- 2 (Active Comparator): Following ethics committee approval, 20 patients with uncontrolled glaucoma will be randomised to trabeculectomy with mitomycin -C. Randomisation is performed. Then, trabeculectomy is performed
  Interventions: Drug: MMC in glaucoma filtering surgery

INTERVENTIONS:
Device: ologen collagen matrix in glaucoma filtering surgery — If ologen™ treatment is used, the collagen matrix will be placed on top of the scleral flap under the conjunctiva after the trabeculectomy.
  Arms: 1
Drug: MMC in glaucoma filtering surgery — If mitomycin -C is applied, a single cellulose sponge soaked with MMC (0.2mg/ml - 0.4mg/ml) is fashioned into an approximate 2.0 × 4.0 mm rectangular shape and applied to the scleral bed and subconjunctival space taking care to avoid exposure to the conjunctival wound edge. Application time is 2 minutes for MMC. Then, the area treated is copiously irrigated with balanced salt solution. After operation, appropriate anti-inflammatory and antibiotic eye-drops will be prescribed.
  Other Names: Mitomycin C
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of the ologen (OculusGen) Biodegradable Collagen Matrix Implant and the MMC group in filtration surgery.

DETAILED DESCRIPTION:
1. Study Objective: To compare the safety and effectiveness of the ologen (OculusGen) Biodegradable Collagen Matrix Implant and the MMC group in filtration surgery. The primary endpoint is to prove the effectiveness via the reduction of IOP, and the secondary endpoint is to prove the safety via the incidence of complications and adverse events.
2. Study Design: The study is designed as an open-label, randomized, parallel, comparative study. Patients who meet the inclusion/exclusion criteria and sign informed consent will be included. After enrollment, patients will be randomized into two groups: trabeculectomy with OculusGen implant or trabeculectomy with mitomycin-C.
3. Follow-Up: There will be 7 post-operative and follow-up visits within 6 months of surgery: postoperative days 1, 7, 14, 30, 60, 90 and 180. A window of ± 7 days is allowed for the 30, 60, 90 day visits and ± 14 days for the 180 day visits. Further follow-up of subjects after the trial will be the responsibility of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over.
* Uncontrolled glaucoma, with failed medical and laser treatment, requiring trabeculectomy.
* Subject able and willing to cooperate with investigation plan.
* Subject able and willing to complete postoperative follow-up requirements.
* Subject willing to sign informed consent form.

Exclusion Criteria:

* Known allergic reaction to mitomycin-C or Bovine collagen.
* Subject is on warfarin and discontinuation is not recommended.
* Normal tension glaucoma.
* Participation in an investigational study during the 30 days preceding trabeculectomy.
* Ocular infection within 14 days prior to trabeculectomy.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
the effectiveness via the reduction of IOP | 180 day

SECONDARY OUTCOMES:
the safety via the incidence of complications and adverse events. | 180 day

CONTACTS AND LOCATIONS:
Overall Officials: Syed Imtiaz Ali, Professor, Principal Investigator — RMC & Allied Hospital
Locations (1):
- RMC & Allied Hospital, Rawalpindi, Punjab Province, Pakistan

REFERENCES:
- [Result] Chen HS, Ritch R, Krupin T, Hsu WC. Control of filtering bleb structure through tissue bioengineering: An animal model. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5310-4. doi: 10.1167/iovs.06-0378. PMID 17122118
- [Result] Hsu WC, Spilker MH, Yannas IV, Rubin PA. Inhibition of conjunctival scarring and contraction by a porous collagen-glycosaminoglycan implant. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2404-11. PMID 10937547
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740